CLINICAL TRIAL: NCT05537688
Title: Identification of Graphic Markers of Neurocognitive Disorders Such as Primary Progressive Aphasia (PPA) and Early-stage Alzheimer's Disease (AD) (MG)
Brief Title: Identification of Graphic Markers of Neurocognitive Disorders (MG)
Acronym: MG
Status: Completed | Type: Observational
Sponsor: Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal (Other Government)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, PhD, Senior researcher, Director of laboratory, Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal
Other Study IDs: 2023-1632
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Alzheimer Disease; Primary Progressive Aphasia; Neurocognitive Disorders
Keywords: Graphic markers
MeSH Terms: conditions — Alzheimer Disease; Aphasia, Primary Progressive; Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: Participants will complete a graphic task included in a validated test for language impairment in adults and the elderly (DTLA).
  They must not have a diagnosis of minor or major neurocognitive disorder.
  Interventions: Behavioral: Identification of Graphic Markers
- Alzheimer's Disease group: Participants will complete a graphic task included in a validated test for language impairment in adults and the elderly (DTLA).
  They must have mild stage Alzheimer's disease: 1/ Be diagnosed according to ICD-10 criteria for the following conditions: Alzheimer's disease and 2/ Have an MMSE score between 20 and 27, corresponding to a major TNC of mild stage or have a diagnosis of minor TNC with an MMSE score between 25 and 30, the validity period of a previously done MMSE is 3 months.
  Interventions: Behavioral: Identification of Graphic Markers
- PPA group: Participants will complete a graphic task included in a validated test for language impairment in adults and the elderly (DTLA).
  They must have Primary Progressive Aphasia according to the Gorno-Tempini criteria (Gorno-Tempini et al., 2011) and have an MMSE score between 20 and 27, corresponding to mild stage major CND or have a diagnosis of minor CND with an MMSE score between 25 and 30, the validity period of a previously made MMSE is 3 months.
  Interventions: Behavioral: Identification of Graphic Markers

INTERVENTIONS:
Behavioral: Identification of Graphic Markers — The study consists of a single physical visit to the research team's site.
  Participants will take a graphic task included in a validated test for language impairment in adults and older adults (DTLA). This test with writing data has a maximum completion time of 15 minutes. Diagnostic data will be collected from the patient's chart, frailty data and socio-demographic data will be collected by self-questionnaires.
  Participants will be evaluated by the principal investigator or his or her representatives from the research team.

SUMMARY:
The diagnosis of neurocognitive disorders such as early Alzheimer's disease (AD) or primary progressive aphasia (PPA) is particularly difficult and constantly evolving, often leading to diagnostic erraticity. However, several studies have shown that graphic parameters are affected in people with moderate to severe Alzheimer's disease. The use of new technologies in the study and analysis of the abilities of people with neurodegenerative diseases is increasingly recommended. The use of a digital tablet with a stylus makes it possible to objectivize the kinematic parameters of writing (pressure, inclination, speed, jerk, time of writing task) and thus would allow a low-cost diffusion of this technology in particular by including it in already existing screening batteries.

The overall objective of the project is to characterize and compare the graphical markers of a writing task, either language-based (writing words, non-words, sentences) or non-language-based (drawing shapes), in patients with PPA, early-stage Alzheimer's disease (i.e., at the stage of minor neurocognitive disorders and major neurocognitive disorders at the beginning of the disease), and in people with no cognitive disorders.

ELIGIBILITY:
Inclusion Criteria:

* = > 50 years old

For control group :

* not have a diagnosis of minor or major neurocognitive disorder.

For AD :

* Have mild stage Alzheimer's disease: 1/ Be diagnosed according to ICD-10 criteria for the following conditions: Alzheimer's disease and 2/ Have an MMSE score between 20 and 27, corresponding to a major TNC of mild stage or have a diagnosis of minor TNC with an MMSE score between 25 and 30, the validity period of a previously done MMSE is 3 months.

For PPA :

* Have Primary Progressive Aphasia according to the Gorno-Tempini criteria (Gorno-Tempini et al., 2011) and have an MMSE score between 20 and 27, corresponding to major mild TNC or have a diagnosis of minor TNC with an MMSE score between 25 and 30, the validity period of a previously made MMSE is 3 months.

Exclusion Criteria:

* Presence of pathologies of the dominant upper limb(s) (left, right or ambidextrous lateralization) disabling such as osteoarthritis, finger amputation, etc.
* History of stroke.
* Illiterate person.
* Participate in a concurrent experimental clinical study, to avoid interference with our study.
* Not understand oral and written French. The speakers are French-speaking and the language task is performed in French.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from the patient files of the principal investigator.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-08-27 (Actual)

PRIMARY OUTCOMES:
Average writing pressure | 3 months
  The primary outcome measure is the difference in writing pressure averages collected between the language and non-language tasks in the three groups of interest.
  It will be assessed using DTLA screening battery (Macoir et al., 2017) to which writing tasks will be added.
Average writing speed | 3 months
  The second primary outcome measure is the difference in writing speed averages collected between the language and non-language tasks in the three groups of interest.
  It will be assessed using DTLA screening battery (Macoir et al., 2017) to which writing tasks will be added.

SECONDARY OUTCOMES:
Physical and autonomy frailty | 3 months
  A physical frailty score will be obtained by using the CARE questionnaire. An autonomy frailty score will be obtained by using ADL and IADL scales.
Socio-demographic characteristics | 3 months
  Participants will be asked their date of birth, sex, gender, lateralization (right-handed, left-handed or ambidextrous), level of education, born in Canada or elsewhere, number of years on Canadian soil, place of living (individual residence, RPP, other), presence of a natural caregiver.
Stage of the neurodegenerative disease | 3 months
  Stage of the neurodegenerative disease will be assessed by using the MMSE test.
  Furthermore, participants will be asked the number of medications taken per day, the use of psychotropic medications (antidepressants, anxiolytics, neuroleptics) and the use of an antidementia treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- CRIUGM, Montreal, Quebec, Canada